CLINICAL TRIAL: NCT03324152
Title: Effects of High-intensity Interval Training (HIIT) Compared to Low-intensity Exercise in Patients With Recent Onset Polymyositis and Dermatomyositis - a Randomized Controlled Trial
Brief Title: Effects of High-intensity Interval Training (HIIT) in Recent Onset Polymyositis and Dermatomyositis
Acronym: HIITmyositis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Helene Alexanderson, Associate professor, RPT, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KarolinskaUH1
Record Dates: First submitted 2017-10-05; First posted 2017-10-27 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Polymyositis; Dermatomyositis
Keywords: High-intensity interval training; Exercise; Muscle function; Inflammation
MeSH Terms: conditions — Polymyositis; Dermatomyositis; Motor Activity; Inflammation | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Patients are dandomized to either a high-intensity interval group (HIIT) or a control group performing standard low-intensity home exercise.
Who Masked: Outcomes Assessor
Masking Description: The physical therapist performing assessments of muscle function (primary outcome), distributes questionnaires and who is present at maximal oxygen uptake tests and who plan all other assessments logistically is blinded to group allocation. The rheumatologists performing assessment of disease activity and the personell analysing biopsy data are also blinded to group allocation. The care provider is the only one who is not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-intensity interval training (HIIT) - myositis (Experimental): 12-week, 3d/w, HIIT
  Interventions: Other: High-intensity interval training (HIIT) - myositis
- Standard low-intensity home exercise control (CG) (Active Comparator): 12-week, 5 d/w, home exercise.
  Interventions: Other: Standard low-intensity home exercise
- High-intensity interval training (HIIT) - healthy (Active Comparator): 12-week, 3d/w, HIIT.
  Interventions: Other: High-intensity interval training (HIIT) - healthy

INTERVENTIONS:
Other: High-intensity interval training (HIIT) - myositis — 12-weeks of 3 days/week HIIT. 6 sets of 30-60 seconds on 85-100% of maximal heart rate performed on a stationary bike followed by resistance training on 10 voluntary repetition maximum.
  Arms: High-intensity interval training (HIIT) - myositis
Other: Standard low-intensity home exercise — 12 weeks of 5 days/week low-intensity resistance home exercise in combination with outdoor walks of 20 minutes.
  Arms: Standard low-intensity home exercise control (CG)
Other: High-intensity interval training (HIIT) - healthy — 12-weeks of 3 days/week HIIT. 6 sets of 30-60 seconds on 85-100% of maximal heart rate performed on a stationary bike followed by resistance training on 10 voluntary repetition maximum.
  Arms: High-intensity interval training (HIIT) - healthy

SUMMARY:
Polymyositis and dermatomyositis are rare inflammatory systemic conditions. Reduced muscle function is a cardinal symptom and lung involvement is very common. Knowledge of heart involvement in these patients is very limited, as is knowledge of exercise effects in recent onset, active disease.

The aim of this project is to investigate effects of high-intensity interval training (HIIT) compared to standard low-intensity home exercise as to tolerance, physical capacity, quality of life, depression, disease activity, inflammation, muscle mass/fat mass, muscle metabolism and heart function in patients with recent onset, active polymyositis and dermatomyositis.

This is a randomized controlled trial. Muscle biopsies are taken at time of diagnosis and after 12 weeks of exercise. Muscle biopsies will be analyzed as to baseline kynurenine pathway, calcium release, gene expression and inflammatory infiltrates and as to changes in these parameters following exercise. Muscle function (primary outcome), maximal oxygen uptake, muscle mass/fat mass, disease activity, systolic and diastolic heart function, as well as quality of life and depression is measured at baseline and after 12 weeks of exercise. After all assessments, patients are randomized to HIIT or standard low-intensity home exercise.

The HIIT group will perform 6 sets of 30-60 second biking bouts reaching 85-100% of maximal heart rate, in combination with strength training, three days a week for 12 weeks. The control group will perform a standardized home exercise program five days a week for 12 weeks. After 12 weeks, all assessments are preformed again. If the HIIT is well tolerated, patients in the control group will be invited to HIIT exercise according to the same protocol. Clinical assessments will be performed at 3, 6 and 9 months follow-up in an open extension.

This study will improve our understanding of heart function, muscle metabolism as well as tolerance and effects of intensive exercise as well as heart function early in the disease course and could also improve treatment and prognosis in patients with polymyositis and dermatomyositis.

DETAILED DESCRIPTION:
Patients randomized to the HIIT protocol will train three days a week for 12 weeks. Before exercise start participants will rate self-reported pain and fatigue on a visual analogue scale and describe in own words information about possible changes in medication dose, any side effects from medication as well as possible negative and positive effects from previous exercise sessions, as well as physical activities performed since the previous exercise session. Each exercise session starts with a 5-minut warm-up on about 50% of maximal heart rate. Each HIIT set is between 30-60 seconds where loads are increased and the participant bikes as fast as possible with the goal of reaching >85% of maximal heart rate. During the 2-minuts rest in-between HIIT sets the participant will rate self-reported exertion using the Borg CR-10, 0-10 scale and the Borg RPE scale, 6-20.

When initiating the exercise period, participants start on three HIIT sets on a lower intensity, gradually increasing to goal intensity during the first two weeks. Then the number of sets are gradually increased to six sets.

After completing six HIIT sets the participants perform one set of 10 voluntary repetitions maximum (VRM) resistance training of the deltoids using free weights and of the quadriceps using free weights or a quadriceps curl machine, depending on degree of muscle weakness. Every other week a new 10 VRM is tested and training loads are adapted. After completing each set, the participant rates perceived muscle exertion on the Borg CR-10 scale. The program is ended with stretching of trained muscle groups and rating of overall exertion during the exercise session on the Borg RPE-scale.

Participants randomized to the control group will perform a standardized home exercise program on an easy-to moderate intensity adapted to initial muscle weakness, five days a week for 12 weeks. The program includes tasks for muscle groups targeted by myositis and takes about 15 minutes to perform. In combination with the home exercise program the participants walks 15 minutes on 60% of maximal heart rate. Participants fill out an exercise diary commenting on loads and number of repetitions for each task.

Participants in both groups ware a Polar 330A heart rate monitor during each training session. By synchronizing to a computer program all exercise data are stored in a cloud data base and can be monitored regularly by the project investigator.

ELIGIBILITY:
Patients with polymyositis and dermatomyositis:

Inclusion Criteria:

* Probable or definite diagnosis polymyositis or dermatomyositis according to Bohand and Peter criteria, diagnosis duration between 4 weeks and 6 months, completed screening for possible concurrent cancer diagnosis and screening for lung involvement, able to performe the HIIT.

Exclusion Criteria:

* Diagnosis of inclusion body myositis, active cancer, being treated for cancer, heart- or lung involvement contraindicating HIIT, no clinical improvement with medical treatment, severe osteoporosis.

Healthy controls:

Inclusion Criteria: match a patient for age and gender, exercising not more than twice a week, no neuro- or musculoskeletal disorders.

Exclusion Criteria: Ongoing treatment for cancer, cardiovascular disease contraindicating a maximal oxygen uptake test or HIIT.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
VO2 max, L/min and ml/kgxmin | 12 weeks
  A maximal oxygen uptake test with ECG on a stationary bike. For patients with myositis, the test is started on 30W and increasing with 10W every minute until exhaustion. Ventilation and gas exchanges is assessed. Definition of max: ration CO2 / O2 = >1. The test is stopped when maximal effort according to above definition is reached or when the subjects cannot bike any longer due to exhaustion. Healthy subjects will start on 50W and then follow the same protocol. Subjects rate subjective exertion of thigh muscles, dyspnea on the Borg symptom scale, 0-10. After completion of test overall exertion is rated on the Borg RPE scale, 6-20.

SECONDARY OUTCOMES:
Aerobic capacity, Watt max | 12 weeks
  A maximal oxygen uptake test with ECG on a stationary bike. For patients with myositis, the test is started on 30W and increasing with 10W every minute until exhaustion. Ventilation and gas exchanges is assessed. Definition of max: ration CO2 / O2 = >1. The test is stopped when maximal effort according to above definition is reached or when the subjects cannot bike any longer due to exhaustion. Healthy subjects will start on 50W and then follow the same protocol. Subjects rate subjective exertion of thigh muscles, dyspnea on the Borg symptom scale, 0-10. After completion of test overall exertion is rated on the Borg RPE scale, 6-20.
Myositis Disease Activity Assessment Tool (MDAAT) - physician's global assessment. | 12 weeks
  A myositis-specific protocol in Biodex systems is used. After completing measures of MVIC, the subjects perform six sets of 12, 4-second contractions with a 6-second rest in-between. Set 1: 12 contractions on 20% of MVIC. For each set, intensity is increased by 10%. In the last, 6th set contractions are performed on 70% of MVIC. After each set, a new MVIC is tested. The MDAAT is a valid core set of measures to assess disease activity including physician's and patient's global assessment, measures of muscle strength, activity limitation and extra-muscular organ activity. Physician's global assessment is performed in a Visual Analogue Scale (VAS), 0-100.
Myositis Disease Activity Assessment Tool (MDAAT) - patient's global assessment | 12 weeks
  The MDAAT Patient's global assessment is performed in a Visual Analogue Scale (VAS), 0-100.
Myositis Disease Activity Assessment Tool (MDAAT) - Manual Muscle Test | 12 weeks
  The MDAAT Manual muscle test measures isometric muscle strength in 8 muscle groups with a composite score varying from 0-80, where 8 indicates good muscle strength.
Myositis Disease Activity Assessment Tool (MDAAT) - Health Assessment Questionnaire (HAQ). | 12 weeks
  The MDAAT, HAQ includes 20 questions about ability to perform daily activities with a composite score varying from 0-3, where 3 indicates severe limitations.
Myositis Disease Activity Assessment Tool (MDAAT) - serum creatine phosphokinase (CK). | 12 weeks
  The MDAAT, serum CK-levels is measured in mikrocat/L.
Myositis Disease Activity Assessment Tool (MDAAT) - MYOACT constitutional | 12 weeks
  The MDAAT, MYOACT constitutional (fever, weight loss) is assessed on a VAS, 0-100.
Myositis Disease Activity Assessment Tool (MDAAT) - MYOACT heart | 12 weeks
  The MDAAT, MYOACT heart involvement is assessed on a VAS, 0-100.
Myositis Disease Activity Assessment Tool (MDAAT) - MYOACT lung | 12 weeks
  The MDAAT, MYOACT lung involvement is assessed on a VAS, 0-100.
Myositis Disease Activity Assessment Tool (MDAAT) - MYOACT skeletal | 12 weeks
  The MDAAT, MYOACT skeletal (joint inflammation and bone density) involvement is assessed on a VAS, 0-100.
Myositis Disease Activity Assessment Tool (MDAAT) - MYOACT gasto-intestinal tract. | 12 weeks
  The MDAAT, MYOACT gastro-intestinal tract involvement such as dysphagia is assessed on a VAS, 0-100.
Myositis Disease Activity Assessment Tool (MDAAT) - MYOACT skin | 12 weeks
  The MDAAT, MYOACT skin involvement (skin rash) is assessed on a VAS, 0-100.
Myositis Damage Index (MDI) - muscle | 6 months
  Degree of skeletal muscle damage is assessed on a VAS, 0-100
Myositis Damage Index (MDI) - lung | 6 months
  Degree of lung dagame is assessed on a VAS, 0-100
Myositis Damage Index (MDI) gastro-intestinal tract | 6 months
  Degree of GI-tract damage is assessed on a VAS, 0-100.
Myositis Damages Index (MDI) Skeletal | 6 months
  Degree of joint damage and osteoporosis is assessed on a VAS, 0-100.
Myositis Damage Index (MDI) heart | 6 months
  Degree of damage of the heart is assessed on a VAS, 0-100.
Stress echocardiography | 12 weeks
  Systolic and diastolic heart function is assessed by ultrasound of the heart.
Inflammatory infiltrates in skeletal muscle | 12 weeks
  Muscle biopsies are analyzed for inflammatory infiltrates with immunohistochemistry.
Gene expression | 12 weeks
  Muscle biopsies are analyzed with Micro Array technique
ER-stress | 12 weeks
  Muscle biopies are analysed by ELIZA
Proteins involved in kynurenine process | 12 weeks
  Muscle biopsies are analyzed by ELIZA
Proteins involved in calcium release | 12 weeks
  Muscle biopsies are analyzed by ELIZA
Isometric muscle strength | 12 weeks
  A myositis-specific protocol in Biodex systems is used. Following several familiarization sets, maximal voluntary isometric contraction (MVIC) is tested until three very similar contractions are recorded. The subjects rest one minute between each MVIC.
Isomteric muscle fatigability | 12 weeks
  A myositis-specific protocol in Biodex systems is used. After completing measures of MVIC, the subjects perform six sets of 12, 4-second contractions with a 6-second rest in-between. Set 1: 12 contractions on 20% of MVIC. For each set, intensity is increased by 10%. In the last, 6th set contractions are performed on 70% of MVIC. After each set, a new MVIC is tested.

CONTACTS AND LOCATIONS:
Overall Officials: Helene Alexanderson, PhD, Ass.Prof, Principal Investigator — Karolinska University Hospital and Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, N/A = Not Applicable, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Muscle biopsies will be sent to Professor Kanneboyina Nagaraju, Professor and Founding Chair, Department of Pharmaceutical sciences, School of Pharmacy and Pharmaceutical Sciences AB-G34, Binghamton University, PO Box 6000 Binghamton, NY 13902-6000. Purpose: To analyse muscle biopsies for micro array analysis.
Supporting Information: Analytic Code
Time Frame: After completion of the project, muscle biopsies from all patients and healthy subjects will be sent to Dr Nagaraju.

REFERENCES:
- [Background] Cleary LC, Crofford LJ, Long D, Charnigo R, Clasey J, Beaman F, Jenkins KA, Fraser N, Srinivas A, Dhaon N, Hanaoka BY. Does computed tomography-based muscle density predict muscle function and health-related quality of life in patients with idiopathic inflammatory myopathies? Arthritis Care Res (Hoboken). 2015 Jul;67(7):1031-40. doi: 10.1002/acr.22557. PMID 25623494
- [Background] Alexanderson H. Physical exercise as a treatment for adult and juvenile myositis. J Intern Med. 2016 Jul;280(1):75-96. doi: 10.1111/joim.12481. Epub 2016 Feb 8. PMID 26854121
- [Background] Yamada T, Place N, Kosterina N, Ostberg T, Zhang SJ, Grundtman C, Erlandsson-Harris H, Lundberg IE, Glenmark B, Bruton JD, Westerblad H. Impaired myofibrillar function in the soleus muscle of mice with collagen-induced arthritis. Arthritis Rheum. 2009 Nov;60(11):3280-9. doi: 10.1002/art.24907. PMID 19877058
- [Background] Yamada T, Fedotovskaya O, Cheng AJ, Cornachione AS, Minozzo FC, Aulin C, Friden C, Turesson C, Andersson DC, Glenmark B, Lundberg IE, Rassier DE, Westerblad H, Lanner JT. Nitrosative modifications of the Ca2+ release complex and actin underlie arthritis-induced muscle weakness. Ann Rheum Dis. 2015 Oct;74(10):1907-14. doi: 10.1136/annrheumdis-2013-205007. Epub 2014 May 22. PMID 24854355
- [Background] Alexanderson H, Munters LA, Dastmalchi M, Loell I, Heimburger M, Opava CH, Lundberg IE. Resistive home exercise in patients with recent-onset polymyositis and dermatomyositis -- a randomized controlled single-blinded study with a 2-year followup. J Rheumatol. 2014 Jun;41(6):1124-32. doi: 10.3899/jrheum.131145. Epub 2014 May 1. PMID 24786930
- [Background] Munters LA, Loell I, Ossipova E, Raouf J, Dastmalchi M, Lindroos E, Chen YW, Esbjornsson M, Korotkova M, Alexanderson H, Nagaraju K, Crofford LJ, Jakobsson PJ, Lundberg IE. Endurance Exercise Improves Molecular Pathways of Aerobic Metabolism in Patients With Myositis. Arthritis Rheumatol. 2016 Jul;68(7):1738-50. doi: 10.1002/art.39624. PMID 26867141
- [Background] Alemo Munters L, Dastmalchi M, Andgren V, Emilson C, Bergegard J, Regardt M, Johansson A, Orefelt Tholander I, Hanna B, Liden M, Esbjornsson M, Alexanderson H. Improvement in health and possible reduction in disease activity using endurance exercise in patients with established polymyositis and dermatomyositis: a multicenter randomized controlled trial with a 1-year open extension followup. Arthritis Care Res (Hoboken). 2013 Dec;65(12):1959-68. doi: 10.1002/acr.22068. PMID 23861241
- [Background] Alemo Munters L, Dastmalchi M, Katz A, Esbjornsson M, Loell I, Hanna B, Liden M, Westerblad H, Lundberg IE, Alexanderson H. Improved exercise performance and increased aerobic capacity after endurance training of patients with stable polymyositis and dermatomyositis. Arthritis Res Ther. 2013 Aug 13;15(4):R83. doi: 10.1186/ar4263. PMID 23941324